CLINICAL TRIAL: NCT03325374
Title: BLB Study Back or Leg Pain and Bladder Symptoms Study
Acronym: BLB
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/NS/0112
Record Dates: First submitted 2017-04-06; First posted 2017-10-30 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cauda Equina Syndrome; Functional Neurological Disorder
MeSH Terms: conditions — Cauda Equina Syndrome; Conversion Disorder | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for genetic storage (DNA) and later study will be requested from all patients. No tests will be done initially. We have an excellent opportunity to better understand the genetics of degenerative disc disease and/or functional disorders using the comparison of DNA between the 'scan positive' and 'scan negative' group.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BLB patients: Patients admitted for urgent MRI with possible cauda equina syndrome will be consented for questionnaires and examination.
  Interventions: Other: Questionnaires and examination

INTERVENTIONS:
Other: Questionnaires and examination — Patients with in the BLB patients study will have interview and questionnaire carried out.

SUMMARY:
The research focuses on Cauda Equina Syndrome (CES) which describes damage to the nerves in the lower back which supply bladder, bowels, sexual function and the legs usually from slipped discs in the spine.

CES is as common as multiple sclerosis and is diagnosed using an MRI scan of the spine, 'scan positive' CES. However, about 50% of people presenting with the symptoms of CES have MRI scans which do not explain their symptoms, 'scan negative' patients. The BLB study will be the first large clinical study comparing patients with 'scan positive' and 'scan negative' CES. All patients admitted to the Western General Hospital, Edinburgh with possible CES will be invited to participate. The study consists of detailed history taking, examination and a questionnaire following up patient's symptoms at three months.

The study aims to see what differences exist between the 'scan positive' and 'scan negative' groups, help doctors understand more about the outcomes of both groups and discover the number of patients with 'scan negative' CES who have functional disorders (previously called medically unexplained or conversion disorders) or undiagnosed neurological disorders.

DETAILED DESCRIPTION:
Uro-neurological disorders are those in which there is a disturbance of bladder function related to a neurological cause. However, many patients with Uro-Neurological disorders are not found to have explanatory abnormalities despite adequate clinical and radiological investigation, so-called 'scan negative' patients. The BLB study will investigate this problem through an acute disorder, Cauda Equina Syndrome (CES), to provide a better understanding of scan-negative Uro-Neurological disorders.

CES is a devastating condition caused by compression of the cauda equina nerve roots resulting in bowel, bladder and sexual dysfunction with potential lower limb weakness. CES requires urgent surgery and has serious potential morbidity and medico-legal consequences1. Suspected acute CES has a minimum incidence of 11 per 100,000 making it twice as common as multiple sclerosis. However, in the two largest studies both retrospective and from Edinburgh, 43-48% of patients with clinical CES were 'scan-negative' and indeed received no other diagnosis 1,2.

Little is known about patients with 'scan negative' CES and nothing is known about their outcome. Our two studies in Edinburgh found basic clinical and demographic characteristics could not distinguish 'scan positive' and 'scan negative' groups 1,2. However, on the basis of clinical experience, and now prospective pilot data, the investigators hypothesise that many of these patients have either an acute functional disorder or, in some cases, sacral nerve damage not seen on imaging but detectable on anal sphincter EMG. Functional disorders, also called psychogenic/non-organic disorders, refer to genuinely experienced physical symptoms which can be positively identified as not related to underlying neurological disease3. Finding out about the diagnosis of patients with 'scan negative' CES would enable them to access treatment and improve their outcome as well as creating better service provision for them in the long term. There is also limited data on long term outcome in patients with 'scan positive' CES and a wish for knowledge from the medical community about what the priorities for patients with 'scan positive' CES are after discharge. The investigators have called the study subsection 'Back or Leg pain with Bladder symptoms' (BLB) study because this most accurately describes the symptoms patients have and we know that describing something negatively to patients (e.g. medically unexplained symptoms)is found by patients to be unhelpful.

The BLB study asks three main questions; do patients with 'scan negative' CES have symptoms of bowel, bladder, sexual dysfunction and lower limb weakness and sensory abnormalities due to a functional disorder?; do a proportion of patients with 'scan negative' CES have missed neurological disease?; what are the outcomes of patients with 'scan negative' and 'scan positive' CES after three months?

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Able to complete online or paper questionnaire.
3. Patients admitted to the regional neurosurgical unit, Western General Hospital, Edinburgh with suspected cauda equina syndrome for an MRI scan. Demographic data from all patients attending any NHS Lothian site who have an MRI scan for suspected CES.

Exclusion Criteria:

1. Age less than 16
2. Inability to communicate (e.g. do not speak English)
3. Inability to complete written or oral surveys or give informed consent
4. Age over 100. The upper age limit is set at 100 to allow the greatest number of participants the opportunity to take part. As the study is a follow up study concerns about mortality and high drop out in this age group led to the upper limit of 100 being set.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 161 participants admitted to the Western General Hospital, Edinburgh with possible CES.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
What proportion of patients with 'scan negative' CES have a functional disorder by clinical consensus. | Nov 15-Aug 18
  Percent of patients with 'scan negative' CES and a functional disorder.

SECONDARY OUTCOMES:
Demographics (age, gender, work status) in patients with 'scan positive' and 'scan negative' CES. | Nov 15-Aug 18
  Demographics
Neurological examination findings, using Medical Research Council (MRC) grading and standardised sensory and reflex examinations in patients with 'scan positive' and 'scan negative' CES. | Nov 15-Aug 18
  MRC grading of strength (0-5, from no power to full power)
Hospital Anxiety and Depression (HADs) scores and Structured clinical interview for DSM (SCID) findings in patients with 'scan positive' and 'scan negative' CES at onset of symptoms and HADs scores three months after symptom onset. | Nov 15-Aug 18
  Hospital Anxiety and Depression (HADs) scores (<8 negative, 8-10 mild, 8-14 moderate, 15-21 severe).
Patient priorities after discharge rated using a visual analogue scale. Options will be pain, bladder symptoms, bowel symptoms, sexual function, sensory disturbance, financial, worry/stress/low mood. | Nov 15-Aug 18
  visual analogue scale from 1 would most value help with to 8 would least value help required
The number of patients with 'scan negative' CES have other neurological disease causing their symptoms. | Nov 15-Aug 18
  Number of patients who have a neurological diagnosis explaining their symptoms at up to one year after discharged with CES symptoms.
The number of patients with 'scan negative' CES who have sacral nerve dysfunction found on EMG. | Nov 15-Aug 18
  with 'scan negative' CES who have sacral nerve dysfunction found on EMG.
Bladder function using Urinary Symptom Profile (USP) in patients with 'scan positive' and 'scan negative' CES at symptom onset and at three months after discharge. | Nov 15-Aug 18
  Urinary Symptom Profile splits symptoms up into stress incontinence(0 none to 9 severe), overactive bladder (0 none to 21 severe), low stream (0 none to nine severe)
Bowel function using The Neurogenic Bowel Dysfunction score in patients with 'scan positive' and 'scan negative' CES at symptom onset and at three months after discharge. | Nov 15-Aug 18
  10-13 is moderate dysfunction, 14 or over is severe dysfunction
Sexual function using the Arizona Sexual Experiences Questionnaire in patients with 'scan positive' and 'scan negative' CES at symptom onset and at three months after discharge. | Nov 15-Aug 18
  Abnormal is >19 or 5 or more on any item or 4 or more on three items

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Hoeritzauer, Principal Investigator — University of Edinburgh
Locations (1):
- Department of Neurosciences, Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No